CLINICAL TRIAL: NCT01182584
Title: Application of Digital Infrared Thermal Imaging in Thyroid Disease and Associated Ophthalmopathy and Dermopathy
Brief Title: Application of Digital Infrared Thermal Imaging (DITI) in Graves' Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan university, National Taiwan university
Other Study IDs: 200811040R
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Graves' Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Graves' disease
- Healthy volunteers

SUMMARY:
Graves' disease is characterized by thyrotoxicosis, goiter, ophthalmopathy and dermopathy. Pathogenesis involves autoimmune process. The investigators think temperatures of the area involved in the inflammation may change. Thus the investigators plan to take temperature pictures of Graves' patients using digital infrared thermal imaging system and observe the change.

DETAILED DESCRIPTION:
We will recruited patients of Graves' disease from out patient clinics. We will perform thyroid echo and soft tissue echo first. Then we let patients sit before the thermal camera and take thermal images of eyes necks and tibia. After data collection, we analyse the relation between temperature and laboratory data such as thyroid function and autoimmune profiles.

ELIGIBILITY:
Inclusion Criteria:

* Graves' disease patients. Healthy people

Exclusion Criteria:

* Pregnancy. <16 years old or > 60 years old

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Graves' disease patients with or without ophthalmopathy and dermopathy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shih, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan